CLINICAL TRIAL: NCT04303091
Title: Assessing the Feasibility and Benefits of a Physical Activity Intervention for Advanced Multiple Myeloma Patients
Brief Title: The Feasibility of a Physical Activity Intervention for Advanced Multiple Myeloma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nicole Culos-Reed (Other)
Responsible Party: Sponsor-Investigator, Dr. Nicole Culos-Reed, Principal Investigator, University of Calgary
Organization: University of Calgary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HREBA.CC-17-0058
Record Dates: First submitted 2019-06-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Multiple Myeloma; Hematologic Neoplasms; Advanced Cancer
Keywords: Physical activity; Exercise; Hematology; Intervention; Supportive cancer care; Multiple myeloma; Resistance training
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single group feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): Single-arm study. Participants enrolled engaged in a 12-week exercise program.
  Interventions: Behavioral: Physical Activity for Advanced Cancer Treatment (PAACT)

INTERVENTIONS:
Behavioral: Physical Activity for Advanced Cancer Treatment (PAACT) — 12-week physical activity intervention. 60 minute group-based exercise classes held once per week. Home-based exercise recommendations provided weekly along with basic take-home exercise equipment. Optional palliative care consultations offered.
  Other Names: PAACT

SUMMARY:
Although physical activity (PA) is commonly used to manage symptoms and enhance quality of life (QOL) in cancer survivors, relatively little is known regarding the benefits in advanced multiple myeloma (MM). The primary aims of the Physical Activity in Advanced Cancer Treatment (PAACT) intervention were to examine (1) program feasibility and (2) potential impact on patient outcomes. It is hypothesized that an exercise intervention will be feasible and potentially impactful.

DETAILED DESCRIPTION:
While the introduction of novel and more effective treatments has seen improved survival in multiple myeloma (MM), the aggressive nature of the disease and these corresponding agents can have a debilitating impact on quality of life (QOL). Exercise can help manage symptoms and enhance QOL in cancer survivors, however relatively little is known regarding the feasibility or benefits of exercise in MM. The purpose of this study was to examine the feasibility of a group- and home-based exercise intervention for individuals with advanced MM. In this single arm study, advanced MM patients (DS stage II-III) participated in a 12-week aerobic and resistance training intervention, with the option of palliative care consultation. Participants attended once weekly supervised group exercise classes and received individually tailored home exercise booklets. Validated measures of physical functioning and patient-reported outcomes, including QOL, fatigue, anxiety, depression, and self-compassion were obtained at baseline and 12-weeks (post-intervention). Optional semi-structured interviews were conducted halfway (week 6) and at the end of the intervention (week 12)

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with advanced (Durie-Salmon stage II-III) multiple myeloma
* 18 years of age or older and given a survival prognosis greater than 6 months
* stable hemoglobin level of ≥80g/L as measured within 2 weeks of enrollment
* no active infections at the time of enrollment.

Exclusion Criteria:

* refusal of informed consent
* geographically inaccessible
* non-English speaking
* co-morbidities that interfere with participation (i.e., severe mobility issues or cognitive impairments)
* known or active history of substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of physical activity program as measured by participant recruitment rate. | 3 months
  Recruitment as defined by the proportion of patients who participate in the study, out of the total number of eligible patients.
Feasibility of physical activity program as measured by attendance of group exercise classes. | 12-weeks
  Attendance is defined by the number of weekly group-exercise classes attended.
Feasibility of physical activity program as measured by attrition rate. | 12-weeks
  Attrition is defined as the number of participants who dropped out of the program after completing the baseline assessment.
Feasibility of physical activity program as measured by safety (as measured by incidence of patient reported adverse events). | 12-weeks
  Safety is described as any adverse event reported by the participants during the 12-week program or fitness assessments, related to program participation.

SECONDARY OUTCOMES:
Change from Baseline Upper Body Muscular Strength (in kilograms) as measured by a grip strength test using a hand dynamometer at 12 weeks. | Baseline (week 0) and 12 weeks
  Total grip strength in kilograms is recorded as the sum from the best score of two trials recorded for each hand. Differences between baseline and post-intervention assessments are evaluated.
Change from Baseline Functional lower body strength (in number of repetitions) as measured by the Chair stand test at 12 weeks. | Baseline (week 0) and 12 weeks
  Chair stand test records the number of times a participant can stand from a seated position in 30 seconds. Differences between baseline and post-intervention assessments are evaluated.
Change from Baseline Lower Body Flexibility (in centimeters) as measured by the Chair Sit and Reach flexibility test at 12 weeks. | Baseline (week 0) and 12 weeks
  In the Chair Sit and Reach Flexibility test, lower body flexibility is assessed by having the participant sit on the edge of a seat. The participant extends the leg being tested in front of the hip, with the heel on the floor and the ankle dorsiflexed approximately 90 degrees. The participant flexes the untested leg so that the sole of the foot is flat on the floor about 6 to 12 inches to the side of the body's midline. With the extended leg as straight as possible and the hands on top of each other (palms down), the participant slowly bends forward at the hip joint, keeping the spine as straight as possible and the head in normal alignment (not tucked) with the spine. The participant reaches down the extended leg, trying to touch the toes, and holds this position for 2 sec. A ruler is ran parallel to the participant's lower leg. Two practice trials are allowed followed by two test trials.The best measurement is taken.
Change from Baseline Upper Body Flexibility (in centimeters) as measured by the Back-Scratch Flexibility test at 12 weeks. | Baseline (week 0) and 12 weeks
  In the Back-Scratch Flexibility test, upper body flexibility is assessed by asking the participant to reach, with the preferred hand (palm down and fingers extended), over the shoulder and down the back while reaching around and up the middle of the back with the other hand (palm up and fingers extended). The participant is allowed two practice trials followed by two test trials.The best measurement is taken.
Change from Baseline Mobility (in seconds) as measured by the 8-foot Timed Up and Go test at 12 weeks. | Baseline (week 0) and 12 weeks
  The 8-foot Timed Up and Go test measures the time to move from a seated position, walk 8 feet, and return to a seated position.The best of two trials is taken.
Change from Baseline Balance (in seconds) as measured by a one-foot balance test at 12 weeks. | Baseline (week 0) and 12 weeks
  Participant's Balance is assessed by measuring the time the participant is able to stand on one-foot. Both feet measured. A 45-second cut-off time is implemented.
Change from Baseline Aerobic Capacity (in meters) as measured by the six-minute walk test at 12 weeks. | Baseline (week 0) and 12 weeks
  In the Six-Minute Walk Test, participants are instructed to walk as far as they can for 6 min around a track. Distances are recorded to the nearest 0.5 m.
Change from Baseline Quality of Life as measured by the The Functional Assessment of Cancer Therapy- Multiple Myeloma (FACT-MM) questionnaire at 12 weeks. | Baseline (week 0) and 12 weeks
  The Functional Assessment of Cancer Therapy- Multiple Myeloma (FACT-MM) questionnaire is comprised of the 27-item FACT-General (FACT-G) scale, which provides information on physical, social, emotional, and functional well-being domains in conjunction with 14 MM-specific supplementary questions. The combined subscales of physical, functional, and MM specific domains contribute to the Trial Outcome Index (TOI) score (range of 0-112). The questionnaire is rated on a 5-point Likert scale, and components can be combined to create a total score, with increases in scores representing improved quality of life.
Change from Baseline Fatigue as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) questionnaire at 12 weeks. | Baseline (week 0) and 12 weeks
  The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) questionnaire is a13-item questionnaire rated on a 5-point Likert scale, and components can be combined to create a total score, with increases in scores representing decreased fatigue.
Changes from Baseline Anxiety as measured by the Hospital Anxiety and Depression Scale (HADs) questionnaire at 12 weeks. | Baseline (week 0) and 12 weeks
  The Hospital Anxiety and Depression Scale (HADs) questionnaire is a 14-item scale. Subscales for anxiety were calculated with a range of 0-21, with low scores (0-7) representing normal levels.
Changes from Baseline Depression as measured by the Hospital Anxiety and Depression Scale (HADs) questionnaire at 12 weeks. | Baseline (week 0) and 12 weeks
  The Hospital Anxiety and Depression Scale (HADs) questionnaire is a 14-item scale. Subscales for depression were calculated with a range of 0-21, with low scores (0-7) representing normal levels.
Changes from Baseline Self-compassion as measured by the Self-Compassion Scale (SCS) at 12-weeks. | Baseline (week 0) and 12 weeks
  The Self-Compassion Scale (SCS) is a 26-item scale. The following subscales are measured on a 5-point Likert scale (1 = almost never to 5= almost always): self- kindness, self-judgment, common humanity, isolation, mindfulness and over-identified items. In this study a grand mean representing an overall measure of self-compassion willl be calculated, with a higher score representing higher levels of self-compassion.
Changes from Baseline Physical Activity Levels as measured by the Godin Leisure Time Exercise Questionnaire (GLTEQ) at 12 weeks. | Baseline (week 0) and 12 weeks
  The Godin Leisure Time Exercise Questionnaire (GLTEQ) assesses current physical activity levels. Participants report on the duration and frequency of mild, moderate, and strenuous PA within a typical week over the past month. Total weekly physical activity is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole r Culos-Reed, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada